CLINICAL TRIAL: NCT00262977
Title: Improving Appropriate Aspirin Use Among Adults With Diabetes in a Primary Care Setting: Using an Electronic Medical Record to Target a Physician-supervised Nurse Practitioner Intervention
Brief Title: Improving Aspirin Use in Diabetes: A Cluster Randomized Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 1402-001
Record Dates: First submitted 2005-12-05; First posted 2005-12-07 (Estimated); Last update posted 2010-07-22 (Estimated); Status verified 2010-07

CONDITIONS: Diabetes Mellitus
Keywords: diabetes mellitus; cardiovascular diseases; aspirin; quality of healthcare
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases

INTERVENTIONS:
Behavioral: Electronic prompt plus patient-directed intervention
Behavioral: Electronic prompt to clinician to prescribe aspirin

SUMMARY:
Our aim is to determine if a patient-directed intervention is more effective than computerized clinician reminders alone for improving aspirin use in adults with diabetes.

DETAILED DESCRIPTION:
Many patients with diabetes do not use aspirin to prevent cardiovascular events. Quality improvement initiatives involving both patients and physicians may be more effective than physician-directed approaches alone.

In a large urban primary care internal medicine practice, this study seeks to test if a patient-directed intervention is more effective than computerized clinician reminders alone for improving the appropriate use of aspirin in adults with diabetes.

The study design is a cluster-randomized trial by physician. The frequency of self-reported regular aspirin use will be compared between patients cared for by physicians in the computerized reminder alone group and the computerized reminder plus physician-supervised, nurse practitioner intervention group.

ELIGIBILITY:
Inclusion Criteria:

Diabetes mellitus

* Age at least 40 years old
* At least 2 clinic visits in the 18 months prior to the intervention

Exclusion Criteria:

* Primary care physician declined enrollment

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2004-09; Study Completion 2005-05

PRIMARY OUTCOMES:
Patient reported aspirin use daily or every other day.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Persell, MD, MPH, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Division of General Internal Medicine, Chicago, Illinois, United States